CLINICAL TRIAL: NCT01608425
Title: Impact Assessment by Introducing Telemedicine Consultations for Treatment of Diabetic Patients With Foot Ulcers in Region of Southern Denmark - Randomized Prospective Study
Brief Title: Ulcer Monitoring in Diabetes Mellitus
Acronym: Telesaar
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johnny Froekjaer (Other)
Collaborators: Region of Southern Denmark (Other); European Commission (Other)
Responsible Party: Sponsor-Investigator, Johnny Froekjaer, Research responsible Chief Surgeon, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Telesaar RH_3
Record Dates: First submitted 2012-05-24; First posted 2012-05-31 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Diabetes Mellitus; Foot Ulcers
Keywords: diabetic foot ulcer; ulcer monitoring; telemedicine consultations; cross-sectoral collaboration
MeSH Terms: conditions — Diabetes Mellitus; Foot Ulcer; Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Control group. Regular treatment.
- Diabetes ulcer monitoring (Experimental): Receives a telemedicine intervention: Diabetes ulcer monitoring.
  Interventions: Procedure: telemedicine consultations

INTERVENTIONS:
Procedure: telemedicine consultations — Replacing 2 out of 3 patient visits to out-patient clinic at hospital with treatment at home from visiting nurse and telemedicine consultations with the specialist doctor.
  Other Names: pleje.net
  Arms: Diabetes ulcer monitoring

SUMMARY:
Telemedicine technology enables a direct and online text- and image communication in the treatment system from patient to the ulcer specialist. The technology is expected to have patient-related, economic and therapeutic benefits. The study is a substudy of a larger project entitled "Renewing Health", where also the economic and management aspects are highlighted. However, only few randomized prospective studies are conducted in this field. The purpose of the study is in a randomized prospective study, to assess the impact of the introduction of the telemedicine technology as consultation form between ulcer-nurses in the primary sector and the wound clinics at the hospitals in the region. It is assessed whether the technology can be adopted without incurring the patient a risk. The study aims to perform an impact analysis of the introduction of new technologies for telemedicine wound monitoring in the treatment of diabetic foot ulcers through different studies.

DETAILED DESCRIPTION:
Through randomized and prospective studies the project will show whether a telemedicine approach to wound care can be used as an alternative to traditional attendance at a wound clinic and document whether this consultation form provides a greater patient-satisfaction and cost savings. The project will document that telemedicine is equivalent to conventional outpatient attendance from a therapeutic aspect in terms of number of hospitalizations, number of extra controls, acute interventions and wound healing.

The project is also investigating the extent of time spent on the personnel side using telemedicine consultations compared with conventional outpatient appearances.

ELIGIBILITY:
Inclusion Criteria:

* Having diabetic foot ulcer
* Referred for out-patient clinic treatment by general practitioner
* Referred for out-patient clinic treatment by a surgical department
* Living in Region of Southern Denmark

Exclusion Criteria:

* Psychiatric disorder
* Dementia
* Chronic alcohol abuse which can affect compliance
* Other disorder then diabetes mellitus that have caused foot ulcer (rheumatoid arthritis or arthritis urica)
* Serious kidney disease which requires dialysis
* Previous foot ulcer - which was part of the study
* Expected healing within 2-4 weeks where only one control (final) is expected

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-06 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Admissions to hospital | from time of inclusion until treatment completed, assessed up to 52 weeks
  The number of admissions, incl, beddays, to hospital relating to ulcer treatment for each randomised patient during the treatment period.
Surgical procedures | from time of inclusion until completed treatment, assessed up to 52 weeks
  The number of surgical procedures (incl. amputations) performed at hospital in realtion to the ulcer during the treatment period.

SECONDARY OUTCOMES:
Ulcer healing | Progress is measured at minimum every 4 weeks during treatment period, assessed up to 52 weeks
  The time from inclusion and start of treatment until ulcer is healed and treatment is stopped.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin S. Rasmussen, MD, Study Director — Odense University Hospital; Johnny Froekjaer, MD, Principal Investigator — Odense University Hospital; Knud B. Yderstraede, MD, Study Chair — Odense University Hospital
Locations (6):
- Denmark (6):
  - South-west Hospital, Esbjerg, Region Syddanmark
  - Lillebaelt Hospital, Kolding, Region Syddanmark
  - Odense University Hospital, Odense, Region Syddanmark
  - Svendborg Hospital, Svendborg, Region Syddanmark
  - Hospital South Jutland, Sønderborg, Region Syddanmark
  - Hospital Lillebaelt, Vejle, Region Syddanmark

REFERENCES:
- [Derived] Fasterholdt I, Gerstrom M, Rasmussen BSB, Yderstraede KB, Kidholm K, Pedersen KM. Cost-effectiveness of telemonitoring of diabetic foot ulcer patients. Health Informatics J. 2018 Sep;24(3):245-258. doi: 10.1177/1460458216663026. Epub 2016 Sep 16. PMID 27638453
- [Derived] Rasmussen BS, Froekjaer J, Bjerregaard MR, Lauritsen J, Hangaard J, Henriksen CW, Halekoh U, Yderstraede KB. A Randomized Controlled Trial Comparing Telemedical and Standard Outpatient Monitoring of Diabetic Foot Ulcers. Diabetes Care. 2015 Sep;38(9):1723-9. doi: 10.2337/dc15-0332. Epub 2015 Jun 26. PMID 26116717